CLINICAL TRIAL: NCT03500211
Title: Lidocaine Patch for Adjunct Analgesia for Postoperative Cesarean Birth Patients
Brief Title: Post-Op Lidocaine Patch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Catherine M Leclair, MD, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 16657
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative
Keywords: Cesarean section; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidoderm; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidoderm 5% Topical Patch (Experimental): 5% lidocaine patch applied at 12 hours after cesarean delivery and removed 24 hours after delivery. A second 5% lidocaine patch applied at 36 hours after cesarean delivery and removed at 48 hours after delivery.
  Interventions: Drug: Lidoderm 5 % Topical Patch
- Sham Topical Patch (Sham Comparator): Sham patch containing no study medication applied at 12 hours after cesarean delivery and removed 24 hours after delivery. A second sham patch containing no study medication applied at 36 hours after cesarean delivery and removed at 48 hours after delivery.
  Interventions: Other: Sham Topical Patch

INTERVENTIONS:
Drug: Lidoderm 5 % Topical Patch — Lidocaine patch after cesarean section delivery.
  Other Names: lidocaine patch
  Arms: Lidoderm 5% Topical Patch
Other: Sham Topical Patch — Sham patch after cesarean section delivery.
  Other Names: sham patch
  Arms: Sham Topical Patch

SUMMARY:
Randomized control trial evaluating use of lidocaine vs placebo patch for post-operative cesarean incision pain.

DETAILED DESCRIPTION:
The purpose of this study is to determine if lidocaine patches decrease post-operative pain associated with cesarean births. While the Lidoderm lidocaine patch has been FDA approved for the treatment of skin pain, it has not been studied in women undergoing cesarean birth who experience postoperative pain. Even though this medication has been used in post-operative pain in published studies, the use of this medicine under these circumstances is still considered experimental. A lidocaine patch may provide added benefit for pain control in addition to standard medicines participants would receive after surgery, such as spinal, intravenous, and oral pain medications following cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients who require a scheduled or non-urgent cesarean birth
* Patient able to receive neuraxial analgesia
* Patient able to give verbal and written consent for both cesarean birth and study

Exclusion Criteria:

* Patients requiring emergent cesarean birth
* Patients allergic to lidocaine or adhesive
* Patients who have already received an epidural during this admission or requiring general anesthesia for cesarean birth
* Patients using chronic oral neuromodulators
* Patients with cardiac disease or using anti-arrhythmic agents
* Patients with fibromyalgia or chronic pain syndromes such as rheumatoid arthritis, osteoarthritis, or lupus.
* Daily narcotic or opiate use for greater than the 2 months prior to enrollment in the study.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Leclair, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (4.0) | 33.7 (5.5) | 33.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 24 | 18 | 42
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (7.7) | 32.3 (8.3) | 32.1 (7.9)
Repeat Cesarean Section [Count of Participants; unit: Participants] | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: 12-hour Postoperative Pain Scores
Description: To determine if lidocaine patch is superior to placebo as an adjunctive therapy for acute postoperative pain. Average pain score in women who have undergone cesarean delivery at 12 hours postoperatively. Measured using a Visual Analog Scale (VAS), a scale which measures pain from 0 to 100 with 0="no pain" and 100="the worst pain you have ever felt".
Time Frame: Postoperative (12 hours)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
Number analyzed (Participants) | 25 | 25
score on a scale | 33.5 (17.0) | 28.8 (21.8)

2. Primary Outcome: 24-hour Postoperative Pain Scores
Description: To determine if lidocaine patch is superior to placebo as an adjunctive therapy for acute postoperative pain. Average pain score in women who have undergone cesarean delivery at 24 hours postoperatively. Measured using a Visual Analog Scale (VAS), a scale which measures pain from 0 to 100 with 0="no pain" and 100="the worst pain you have ever felt".
Time Frame: Postoperative (24 hours)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
Number analyzed (Participants) | 25 | 25
score on a scale | 34.1 (23.1) | 32.9 (20.0)

3. Primary Outcome: 36-hour Postoperative Pain Scores
Description: To determine if lidocaine patch is superior to placebo as an adjunctive therapy for acute postoperative pain. Average pain score in women who have undergone cesarean delivery at 36 hours postoperatively. Measured using a Visual Analog Scale (VAS), a scale which measures pain from 0 to 100 with 0="no pain" and 100="the worst pain you have ever felt".
Time Frame: Postoperative (36 hours)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
Number analyzed (Participants) | 24 | 24
score on a scale | 37.3 (13.4) | 43.0 (22.8)

4. Primary Outcome: 48-hour Postoperative Pain Scores
Description: To determine if lidocaine patch is superior to placebo as an adjunctive therapy for acute postoperative pain. Average pain score in women who have undergone cesarean delivery at 48 hours postoperatively. Measured using a Visual Analog Scale (VAS), a scale which measures pain from 0 to 100 with 0="no pain" and 100="the worst pain you have ever felt".
Time Frame: Postoperative (48 hours)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
Number analyzed (Participants) | 24 | 24
score on a scale | 24.8 (16.1) | 29.6 (23.6)

5. Secondary Outcome: 5-days Postoperative Narcotic Use
Description: To determine if narcotic use changes when patients use lidocaine patches by counting amount and frequency of narcotic use over admission. Average number of 5 mg oxycodone pills used in women who have undergone cesarean delivery assessed through questionnaire at 5 days postoperatively.
Time Frame: Postoperative (5 days)
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
Number analyzed (Participants) | 24 | 25
pills | 8.6 (4.4) | 8.3 (5.2)

ADVERSE EVENTS:
Time Frame: Up to 5 days post-operation
Arm/Group | Lidoderm 5% Topical Patch | Sham Topical Patch
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03500211/Prot_SAP_000.pdf